CLINICAL TRIAL: NCT04717284
Title: A Self-compassion Intervention for Parents of Children With Inflammatory Bowel Disease (IBD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sheffield (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 169973
Record Dates: First submitted 2020-12-07; First posted 2021-01-22 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2021-04

CONDITIONS: Inflammatory Bowel Diseases
Keywords: Self-compassion; Parental support; Inflammatory Bowel Disease
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-compassion intervention (SCI) (Experimental): Self-compassion prompt.
  Interventions: Other: Self-compassion intervention (SCI)
- Control condition (Other): Neutral prompt during the initial administration and no intervention during the two-week follow-up.
  Interventions: Other: Control condition

INTERVENTIONS:
Other: Self-compassion intervention (SCI) — All participants will be asked to recall a recent parenting event they feel ashamed of and type it into a text box provided. Participants in the SCI group will then be instructed to reflect on their recalled parenting event and prompted to think about and write about the event in a self-compassionate manner. The prompt is designed to induce on all of the three key elements of self-compassion described by Neff (2003a): self-kindness; common humanity; and mindfulness. The same instructions will be provided for follow-up period.
  Arms: Self-compassion intervention (SCI)
Other: Control condition — All participants will be asked to recall a recent parenting event they feel ashamed of and type it into a text box provided. Participants in the control group will then be instructed to make notes about factual information of the event (e.g. time of day, who was there, the weather, etc.). During the two-week follow-up period, participants in the control group will not take part in any intervention as part of the trial.
  Arms: Control condition

SUMMARY:
Parenting a child with Inflammatory Bowel Disease (IBD) can understandably be challenging and distressing at times. The aim of this study is therefore to investigate the effectiveness of an online self-compassion intervention (SCI), that focuses on helping individuals respond to themselves in a kinder and more accepting way, for parents of children with IBD.

Around 150 parents of children with IBD will be randomly allocated to receive either the online SCI or a control condition. This will involve an initial administration and a two-week follow-up period. Participants will complete outcome measures of self-compassion, distress and shame at three time points.

We hypothesise that, in comparison to a control group, participants receiving the online SCI will: (1) report increased state self-compassion and reduced state shame and distress immediately following the SCI; and (2) report increased trait self-compassion and reduced parental stress after repeated engagement in the SCI materials for two weeks.

Through understanding the effectiveness of an online SCI for parents of children with IBD, we hope that our research will help to inform and improve parental support offered to parents of children with IBD.

DETAILED DESCRIPTION:
INTRODUCTION:

Inflammatory Bowel Disease (IBD) is a diagnostic term encompassing Crohn's disease (CD) and ulcerative colitis (UC), chronic health conditions (CHCs) characterised by parts of the gut becoming swollen, inflamed and ulcerated. Children with IBD are likely to depend on the support of others, particularly their parents and carers.

Parenting a child with a CHC, such as IBD, has been related to feelings of shame and distress in the literature. Despite this, gaps have been identified in the support offered to parents of children with IBD.

When considering how to target the distress associated with parenting a child with IBD, research suggests that self-compassion interventions may be of particular significance. Despite this, no study to our knowledge has explored the benefits of self-compassion for parents of children with IBD.

The current study therefore aims to investigate the effectiveness of an online self-compassion intervention (SCI) for parents of children with IBD.

AIMS:

Primary Aim: To determine the effectiveness of an online SCI in increasing state self-compassion and reducing state shame and distress in parents of children with IBD.

Secondary Aim: To determine the effectiveness of repeated engagement in the SCI materials in increasing trait self-compassion and reducing parental stress in parents of children with IBD.

HYPOTHESES:

Primary Hypotheses: In comparison to a control group, participants receiving the SCI will: 1) report increased state self-compassion immediately following the SCI; 2) report reduced state shame immediately following the SCI; 3) report reduced state distress immediately following the SCI.

Secondary Hypotheses: In comparison to a control group, participants receiving the SCI will: 4) report increased trait self-compassion after repeated engagement in the SCI materials for two weeks; 5) report reduced parental stress after repeated engagement in the SCI materials for two weeks.

METHODS:

DESIGN: See 'Study Design' for information.

PUBLIC AND PATIENT INVOLVEMENT (PPI): Consultation regarding the suitability and feasibility of the design, outcome measures and materials used for this study has been sought through Crohn's and Colitis UK' s (CCUK) virtual PPI in research day.

PARTICIPANTS: A priori power analysis was conducted using G*Power 3. This analysis indicated that it would be necessary to recruit 128 participants in total (64 in each condition) in order to detect a medium effect size, with 80% power and a critical p-value of .05. A medium effect size was predicted as a previous similar study found medium to large effect sizes across their results. The power and critical significance levels were set at 0.8 and 0.05 respectively as recommended in psychological research. The target participant number has been inflated by 20% to account for attrition, this means that we will need to recruit 154 participants in total (77 per group). See Enrolment and Eligibility for more participant information.

DATA COLLECTION AND PROCEDURE: Participants will access a Qualtrics® link which will first ask them to read an information sheet, confirm their informed consent and answer a screening question to determine eligibility.

Participants will then be asked to complete a brief demographic questionnaire along with baseline (Time 1 [T1]) measures of state self-compassion, state shame, state distress, trait self-compassion and parental stress (presented in a randomised order). Participants will then be asked to recall a recent parenting event they feel ashamed of and type it into a text box. A one-item question will then be administered to assess whether feelings of shame have been elicited by the recall task. The randomiser tool on Qualtrics® will then be used to allocate participants to either a control condition or the SCI (see 'Arms, Groups and Intervention' for more information.). After this initial administration, participants will be asked to complete post-condition (Time 2 [T2]) measures of state self-compassion, state shame and state distress to assess for any immediate changes. All participants will then be asked to complete a mood neutralisation task used in previous research to neutralise any potential distress experienced through participation.

Participants in the SCI group will then be asked to engage in the SCI condition every-day for two-weeks. Qualtrics® will be pre-programmed to send participants in this group a daily reminder email during this time which will include a link to a Qualtrics® page containing the instructions and space to engage in the SCI. Participants in the control group will be told they do not need to do anything for two-weeks. After two weeks, Qualtrics® will be pre-programmed to email participants with a link for them to complete follow-up (Time 3 [T3]) measures of trait self-compassion and parental stress. Participants in the SCI group will also be presented with a single item to assess participants' adherence to their allocated condition (e.g. 'how often did you engage in the task? every day [14 days), most days [10-13 days], some of the days [5-9 days], not many of the days [1-4 days], none of the days [0 days]').

All participants will then be presented with a debrief information sheet and information on how to access and continue engaging in the SCI materials.

See 'Arms, Groups and Intervention' for more information.

OUTCOME MEASURES: See 'Outcome Measures' for information

DATA SECURITY: A Data Management Plan (DMP) has been completed in accordance with the University of Sheffield's Research Data Management Policy. The DMP describes the data that will be collected and how it will be managed both during and after the research.

PROPOSED DATA ANALYSIS: Preliminary Analysis: Screening, recruitment, random allocation and treatment engagement (including dropout) data will be summarised using a CONSORT diagram. Appropriate descriptive statistics will be reported. Tests to check for necessary assumptions; differences between groups at baseline; and differences between completers and non-completers will also be conducted and reported, with appropriate adjustments made to the following statistical analysis if necessary. A regression analysis will also be conducted to identify any additional predictors of change (e.g. demographic variables, T1 scores) in each of the dependent variables (DV)s at T2 and T3.

Statistical Analysis:

Hypothesis 1: State self-compassion scores at T2 will be compared using a one-way independent ANCOVA, with condition (SCI or control group) as the between groups independent variable (IV). State self-compassion scores at T1 will be included as a covariate, as recommended for pre-post designs assessing for an intervention effect (Field, 2005). As it has been suggested that research exploring SCIs should control for individual differences in self-compassion, baseline trait self-compassion scores will therefore be included as a covariate, along with any other demographic variables or T1 scores that predicted change in this DV at T2.

Hypothesis 2: State shame scores at T2 will be compared using a one-way independent ANCOVA, with condition (SCI or control group) as the between groups IV. As above, state shame scores at T1, as well as trait self-compassion and any other related variables, will be included as covariates.

Hypothesis 3: State distress scores at T2 will be compared using a one-way independent ANCOVA, with condition (SCI or control group) as the between groups IV. As above, state distress scores at T1, as well as trait self-compassion and any other related variables, will be included as covariates Hypothesis 4: Trait self-compassion scores at T3 will be compared using a one-way independent ANCOVA, with condition (SCI or control group) as the between groups IV. As above, trait self-compassion scores at T1, as well as any other related variables, will be included as covariates.

Hypothesis 5: Parental distress scores at T3 will be compared using a one-way independent ANCOVA, with condition (SCI or active-control group) as the between groups IV. As above, parental distress scores at T1, as well as trait self-compassion and any other related variables, will be included as covariates.

*Both intention-to-treat analysis (including all randomised participants) and per-protocol analysis (only participants who indicate they have engaged in their allocated task for ≥ some of the days [5-9 days]) will be ran to enhance interpretations.

ELIGIBILITY:
Inclusion Criteria:

* Parental responsibility stated.
* Children must be under 18 years old and residing with the parent.
* Children must be diagnosed with IBD.

Exclusion Criteria:

- Not able to read and write in English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2021-04-20 (Actual); Primary Completion 2021-12-11 (Actual); Study Completion 2021-12-11 (Actual)

PRIMARY OUTCOMES:
State self-compassion. | Immediately after the initial administration of the self-compassion intervention (SCI) or control condition (Time 2).
  Five items developed and used by a similar study based on previous research will be used to assess state self-compassion. Participants will use a 7-point Likert scale to rate how they feel 'right now' on items corresponding to the three components of self-compassion: self-kindness; common humanity; and mindfulness. A total score is generated by reversing negative items and calculating a mean of all item scores. The minimum score is 1 and the maximum score is 7. A higher total score indicates greater state self-compassion.
State shame and distress. | Immediately after the initial administration of the self-compassion intervention (SCI) or control condition (Time 2).
  Fourteen items from the Positive and Negative Affect Schedule Expanded Form (PANAS-X) that make up two subscales of guilt and negative affect will be used to assess state shame and distress respectively. Participants will be asked to use a 5-point Likert scale to rate what extent they are experiencing feelings related to shame and distress 'right now (that is, at the present moment)'. A total score for each subscale is calculated by summing the relevant item responses, with higher scores on each subscale indicating greater state shame and distress respectively. The guilt subscale used to assess state shame yields a minimum score of 6 and a maximum score of 30. The negative affect subscale used to assess distress yields a minimum score of 10 and a maximum score of 50.

SECONDARY OUTCOMES:
Trait self-compassion. | After repeated engagement in the self-compassion intervention (SCI) or nothing for the control group for two weeks (Time 3).
  The 26-item Self-Compassion Scale (SCS) will be used to assess parent's trait self-compassion. Participants will use a 5-point Likert scale to rate how often they respond in different ways to assess each of the dimensions of self-compassion. Six subscale scores based on each of the dimensions are computed by calculating the mean of relevant item responses. A total score is generated by reversing negative items and calculating a mean of all six subscale means. The total and subscale scores will be a minimum of 1 and a maximum of 5. Higher total and subscale scores indicate greater trait self-compassion.
Parental stress. | After repeated engagement in the self-compassion intervention (SCI) or nothing for the control group for two weeks (Time 3).
  The Pediatric Inventory for Parents (PIP) will be used to assess parental stress. Participants will use a 5-point Likert scale to rate both the frequency and difficulty of 42 items related to caring for children with CHCs. The measure generates separate scores of stress frequency (F) and difficulty (D) across four domains: Communication; Medical Care; Role Functioning; and Emotional Distress, as well as total frequency (Total-F) and total difficulty (Total-D) scores. For the Total-F and Total-D, the minimum score is 42 and the maximum score is 210. In all cases, higher scores indicate greater illness-related parental stress.

CONTACTS AND LOCATIONS:
Overall Officials: A Wray, Principal Investigator — University of Sheffield
Locations (1):
- Clinical Psychology Unit, University of Sheffield, Sheffield, South Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Anonymous survey data will be deposited in Online Research Data (ORDA; the University of Sheffield data repository), Unidrive (shared drive that has limited access - myself, Research Support Officer, certain members of Psychology department), and an open access data repository (if a condition to publication specified by a journal). Participants will be asked to provide consent for their anonymous survey data to be shared in this way.
Time Frame: Data to be deposited in ORDA and Unidrive after completion of the research project (by September 2022). This will be temporarily embargoed, until the research has been published. Whilst embargoed, contact details will be provided for others to request access if appropriate.
Access Criteria: Whilst data is embargoed prior to publication, contact details will be provided for others to request access if appropriate. Following publication, access to this data will not be restricted.

REFERENCES:
- [Background] Sirois FM, Bogels S, Emerson LM. Self-compassion Improves Parental Well-being in Response to Challenging Parenting Events. J Psychol. 2019;153(3):327-341. doi: 10.1080/00223980.2018.1523123. Epub 2018 Oct 30. PMID 30376651
- [Background] Watson, D., & Clark, L. A. (1994). The PANAS-X: Manual for the positive and negative affect schedule - expanded form. The University of Iowa. https://www2.psychology.uiowa.edu/faculty/clark/panas-x.pdf
- [Background] Breines JG, Chen S. Self-compassion increases self-improvement motivation. Pers Soc Psychol Bull. 2012 Sep;38(9):1133-43. doi: 10.1177/0146167212445599. Epub 2012 May 29. PMID 22645164
- [Background] Neff, K. D. (2003). The development and validation of a scale to measure self-compassion. Self and Identity, 2(3), 223-250. https://doi.org/10.1080/15298860309027
- [Background] Streisand R, Braniecki S, Tercyak KP, Kazak AE. Childhood illness-related parenting stress: the pediatric inventory for parents. J Pediatr Psychol. 2001 Apr-May;26(3):155-62. doi: 10.1093/jpepsy/26.3.155. PMID 11259517
- [Background] Neff, K. D. (2003). Self-compassion: An alternative conceptualization of a healthy attitude toward oneself. Self and Identity, 2(2), 85-101. https://doi.org/10.1080/15298860309032